CLINICAL TRIAL: NCT01145144
Title: Dehydroepiandrosterone Supplementation for Poor Responder Patients During in Vitro Fertilization Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Adriam Shulman, IVF Unit Meir Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mmc07204-2006ctil
Record Dates: First submitted 2010-05-03; First posted 2010-06-16 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Ovarian Stimulation
Keywords: Dehydroepiandrosterone; DHEA; IVF outcome; long protocol IVF; poor-responder; recombinant LH; embryo quality; pregnancy rate; live birth rate; poor response to ovarian stimulation

ARMS (2):
- DHEA supplementation (Experimental): DHEA was added to induction of ovulation by recombinant FSH and recombinant LH, in IVF long protocol
  Interventions: Drug: dehydroepiandrosterone crystalline fine powder
- only induction of ovulation by same long protocol without DHEA (No Intervention)

INTERVENTIONS:
Drug: dehydroepiandrosterone crystalline fine powder
  Arms: DHEA supplementation

SUMMARY:
The aim of this study was to evaluate the effect of dehydroepiandrosterone supplementation on in vitro fertilization performance and outcome among poor-responder patient.

ELIGIBILITY:
Inclusion Criteria:

* previous poor response to ovarian stimulation in IVF.

Exclusion Criteria:

* patients over the age of 42
* patients who received DHEA at any time.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
peak estradiol level.
number of retrieved oocytes.
Embryos that were graded as a top quality (according to the number of cells and percent of fragmentation)
number of embryos reserved for transfer.

SECONDARY OUTCOMES:
pregnancy rate.
live birth rate.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Meir Medical center IVF unit, Kfar Saba, Kfar Saba
  - Meir Medical Center, Kfar Saba, Kfar Sava

REFERENCES:
- [Derived] Wiser A, Gonen O, Ghetler Y, Shavit T, Berkovitz A, Shulman A. Addition of dehydroepiandrosterone (DHEA) for poor-responder patients before and during IVF treatment improves the pregnancy rate: a randomized prospective study. Hum Reprod. 2010 Oct;25(10):2496-500. doi: 10.1093/humrep/deq220. Epub 2010 Aug 21. PMID 20729538